CLINICAL TRIAL: NCT05504317
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AK111 in Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: A Study of AK111 in Subjects With Moderate-to-severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK111-102
Record Dates: First submitted 2022-06-29; First posted 2022-08-17 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK111 regimen (Experimental)
  Interventions: Drug: AK111
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK111 — Subjects will receive one of four escalated doses of AK111 (75mg/150mg/300mg/450mg) injection subcutaneously.
  Arms: AK111 regimen
Drug: Placebo — Subjects will receive corresponding dose of placebo injection subcutaneously.
  Arms: Placebo

SUMMARY:
This is a Phase Ib clinical study of multiple dose escalation of AK111 in subjects with moderate-to-severe plaque psoriasis

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase Ib clinical study. This study aims to determine the safety, tolerance, pharmacokinetics(PK) and Pharmacodynamics (PD) characteristics, immunogenicity and preliminary clinical efficacy of multiple dose escalation administration of AK111 in subjects with moderate-to-severe plaque psoriasis..

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe plaque-type psoriasis diagnosed for at least 6 months;
2. Subjects with moderate-to-severe plaque psoriasis at baseline, who were defined as follows: Body Surface Area (BSA) ≥ 10%, PASI ≥ 12 and SPGA score ≥ 3;
3. Subjects with a history of systemic therapy or phototherapy for psoriasis at least once before, or suitable to receive systemic therapy or phototherapy for psoriasis assessed by investigator;
4. Women of childbearing age is not pregnant or lactating, and the subjects and their partners voluntarily take contraceptive measures considered effective by the investigator during the treatment period and at least 6 months after the last receipt of the study drug.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type psoriasis;
2. History or evidence of active/latent tuberculosis;
3. Positive results of confirmatory serology test for hepatitis B, hepatitis C,HIV or syphilis at screening;
4. History of serious infection within 2 months before screening;
5. History of malignancy of any organ system;
6. Inadequate washout period for prior psoriatic therapy;
7. Previous use of secukinumab, ixekizumab or any other drug that targets IL-17 or IL-17 receptor;
8. Any medical conditions, in the opinion of the investigator, would place the subject at risk, interfere with study participation or study results interpretation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety | Baseline till Week 20
  Incidence of treatment emergent adverse events (TEAE), serious adverse events (SAE).
PK evaluation: T1/2 | Baseline till week 20
  Assessment of elimination half-life (T1/2) after AK111 administration.
PK evaluation: AUC | Baseline till week 20
  Assessment of area under curve (AUC) after AK111 administration.
PK evaluation: Cmax | Baseline till week 20
  Assessment of maximum plasma concentration (Cmax) after AK111 administration.
PK evaluation: Tmax | Baseline till week 20
  Assessment of time to maximum plasma concentration (Tmax) after AK111 administration.

SECONDARY OUTCOMES:
PASI 75 | At week 12
  Proportion of subjects who achieve Psoriasis Area and Severity Index (PASI) 75 response which means whose PASI score decrease at least 75 percent compared with baseline at week 12.
  PASI is a measure of overall psoriasis severity and coverage. The PASI score is in the range of 0 (no psoriasis on the body) to 72 (the most severe case of psoriasis).
PASI 90 | At week 12
  Proportion of subjects who achieve PASI 90 response which means whose PASI score decrease at least 90 percent compared with baseline at week 12.
  PASI is a measure of overall psoriasis severity and coverage. The PASI score is in the range of 0 (no psoriasis on the body) to 72 (the most severe case of psoriasis).
PASI 100 | At week 12
  Proportion of subjects who achieve PASI 100 response which means whose PASI score decrease 100 percent compared with baseline at week 12.
  PASI is a measure of overall psoriasis severity and coverage. The PASI score is in the range of 0 (no psoriasis on the body) to 72 (the most severe case of psoriasis).
sPGA 0/1 | At week 12
  Proportion of subjects who achieve Static Physicians Global Assessment (sPGA) 0/1 which means whose sPGA score is clear or almost-clear at week 12.
  The sPGA is a measure of global assessment of the patient's overall severity, which could be converted to numerals ranging from 0 to 5 (clear = 0, almost-clear = 1, mild = 2, moderate = 3, marked = 4, and severe = 5).
Immunogenicity | Baseline till week 20
  Proportion of subjects with detectable anti-drug antibody (ADA).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - AkesoBio Investigative Site 1002, Bengbu, Anhui
  - AkesoBio Investigative Site 1001, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang C, Zhou H, Zhang W, Xia Y, Li B, Ni X, Wang G, Zhang W, Chen B, He Z, Zhang M, Chen R, Jin H, Deng L. Efficacy, Safety and Pharmacokinetics of IL-17 Monoclonal Antibody Injection (AK111) in Patients with Moderate-to-Severe Plaque Psoriasis: A Randomized, Double-Blinded, Placebo-Controlled Phase Ib Multidose Escalation Clinical Study. Dermatol Ther (Heidelb). 2023 Feb;13(2):555-567. doi: 10.1007/s13555-022-00880-1. Epub 2022 Dec 24. PMID 36566344